CLINICAL TRIAL: NCT01041261
Title: Randomized, Pilot Study to Compare the Effects of a Novel Dietary Intervention With the Post-operative Standard of Care on Body Composition After Laparoscopic Gastric Bypass Surgery
Brief Title: Effects of a Novel Dietary Intervention on Body Composition After Laparoscopic Gastric Bypass Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: MetaProteomics LLC (Industry)
Collaborators: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BAR1-BMC-CT
Record Dates: First submitted 2009-12-29; First posted 2009-12-31 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Obesity; Morbid Obesity
Keywords: Laparoscopic gastric bypass surgery; Medical food; Body composition; Dietary intervention
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (No Intervention): Subjects will be issued control study product (Carnation Instant Breakfast, no sugar added)
- Treatment arm (Experimental): Medical food
  Interventions: Dietary Supplement: BariatrX Essentials 360 Treatment

INTERVENTIONS:
Dietary Supplement: BariatrX Essentials 360 Treatment — Medical food
  Other Names: BariatrX Essentials 360
  Arms: Treatment arm

SUMMARY:
We propose to compare the standard of care with the use of a novel medical food in 6 bariatric surgery patients by measuring outcomes of body composition, quality of life, hair loss, muscle strength, resting energy expenditure, and biochemical parameters.

DETAILED DESCRIPTION:
STUDY SUMMARY The purpose of this pilot study is to compare a medical food intervention with the dietary standard of care at Boston Medical Center, in obese women subjects undergoing Roux-en Y gastric bypass surgery. Commercially available nutritional supplements will also be provided as part of the study's protocol.

Subjects will be selected from surgical candidates of the Nutrition and Weight Management Center who meet the study criteria. Subjects will be randomly assigned to one of the 2 groups (treatment and control). Subjects will be seen at the study site 2 weeks before surgery and 4 weeks, 8 weeks, 12 weeks, and 6 months after surgery (for a total of 5 visits). Data recorded during the study visits will be used to assess post-operative progress and will include: body composition, resting energy expenditure, muscle strength, quality of life questionnaires, hair loss, and blood markers for insulin resistance, nutritional state, organ function, lipid profile and inflammation. Safety indicators and compliance will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Obese and morbidly obese women (BMI 30 - 50)
* 25 years and older undergoing laparoscopic gastric bypass surgery
* Present with at least either metabolic syndrome or diabetes

Exclusion Criteria:

* Have smoked in the past 4 weeks
* Pregnant
* Allergic or intolerant to ingredients used in the study (e.g. soy and THIAA)
* There is a sound medical, psychiatric and/or social reason as determined by the Principal Investigator (PI) that makes the subject unsuitable for the study

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Total and extracellular water (by cold bromide and deuterium method) | Baseline, 4 weeks, 12 weeks, and 24 weeks post surgery
Dual energy X-ray absorptiometry (DEXA) | Baseline, 4 weeks, 12 weeks, and 24 weeks post surgery

SECONDARY OUTCOMES:
Hair loss (by photographic method and Hair-Scalp Questionnaire) | Baseline, 12 weeks, and 24 weeks
Impedance plethysmography (by distal and proximal electrode placement) | Baseline, 4 weeks, 8 weeks, 12 weeks, and 24 weeks
Muscle strength (by a handgrip dynamometer) | Baseline, 4weeks, 12 weeks, and 24 weeks
Resting energy expenditure (by indirect calorimetry) | Baseline, 4 weeks, 12 weeks and 24 weeks
Pulse after a 6-minute walk | Baseline, 4 weeks, 12 weeks, and 24 weeks
Measures of insulin resistance, visceral protein/nutritional status, and inflammation | Baseline, 12 weeks, and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Apovian, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States